CLINICAL TRIAL: NCT00453024
Title: Anterior Segment Optical Coherence Tomography Findings in Patients With Ahmed Glaucoma Drainage Implants With Either a Pericardial Patch Graft and Fibrin Tissue Glue or a Partial-Thickness Scleral Flap and Conventional Sutures
Brief Title: Imaging Ahmed Glaucoma Tubes With a Pericardial Graft and Tissue Glue or Partial-Thickness Scleral Flap and Sutures
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Cecilia Aquino, MD
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSRB A/06/375
Record Dates: First submitted 2007-03-27; First posted 2007-03-28 (Estimated); Last update posted 2008-05-14 (Estimated); Status verified 2008-05

CONDITIONS: Advanced Glaucoma; Failed Trabeculectomies
Keywords: Advanced glaucoma; Ahmed glaucoma implant; Anterior segment optical coherence tomography; Pericardial patch graft; Tissue glue; Scleral flap; Sutures
MeSH Terms: interventions — Sutures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Pericardial graft & tissue glue
Procedure: scleral flap & sutures

SUMMARY:
When implanting an Ahmed glaucoma tube, a scleral flap is usually created to cover the tube, and the conjunctiva is stitched back in place with nylon 10-0 sutures. It is hypothesized that an equally safe or better method is using a bovine pericardial patch graft that can be secured in place over the tube with tissue glue, and using tissue glue to reposition the conjunctiva in place.

DETAILED DESCRIPTION:
Glaucoma drainage devices (GDD) are usually reserved for cases wherein filtration surgery has failed, or for difficult cases that do not respond to filtration surgery, such as neovascular or uveitic glaucoma.

The Ahmed Glaucoma drainage implant (New World Medical, Rancho, Cucamonga,CA) was introduced to the market in 19942. It has a scarab-shaped end plate made of polypropylene (models S2, S3 and B1) or silicone models (FP7, FP8 and FX1). Fenestrations have been added to the end plate of the silicone models. Various sizes of the Ahmed drainage are available, including those with a surface area of 96 mm2 (S3 and FP8) or 184 mm2 (S2 and FP7); while the double-plate version has a surface area of 364mm2 (B1 and FX1). Aqueous humor passes from the anterior chamber through two thin membrane-like elastomer sheets that theoretically restrict flow until a pressure of greater than 8-12 mm Hg is exerted on them.

In the implantation of GDD, absorbable and non-absorbable sutures are used. Sutures are typically used in securing the plate to the sclera, securing the tube to the sclera, suturing a patch graft or scleral flap over the silicone tube, and for conjunctival closure. Post-surgical course can be marked by discomfort, depending on the type of suture used. Absorbable sutures can induce inflammation with localized surface and subconjunctival fibrosis that leads to uneven conjunctival surface and excessive scarring. On the other hand, non-absorbable sutures can erode through tissue post-operatively. Suturing the conjunctiva can cause button-holes and tears, and can be the most time-intensive portion of the surgery.

Fibrin glue has been used in various ophthalmic surgeries such as a sealant for perforated and preperforated corneal ulcers, in mucous membrane grafts, in the management of complicated hypotony and bleb leaks after trabeculectomy, and for preventing immediate postoperative hypotony after glaucoma drainage implant surgery.

In a paper by Kahook and Noecker published in 2006, the authors did a retrospective non-randomized case-control study that reviewed 28 cases of GDD implantations using traditional suture materials compared to 14 consecutive cases of GDD implantation using Tisseel fibrin glue (Baxter AG, Vienna, Austria) for closing the conjunctiva, securing the pericardium patch graft and securing the tube to the sclera. The authors concluded that Tisseel fibrin glue seems to be a safe substitute for some of the sutures used in GDD surgery; and it has no impact on IOP control or complications. It appears to reduce post-operative conjunctival inflammation and time of surgery.

Optical coherence tomography (OCT) is a high-resolution, non-invasive and reproducible imaging technology that was primarily developed to evaluate the retina and retina nerve fiber layer in patients with vitreo-retinal or optic nerve diseases11. Recently, the anterior segment OCT (AS-OCT) has been developed and used to image anterior segment structures. It has also been used to localize the Ex-PRESS miniature glaucoma implant in porcine eyes, while the conventional OCT was used to show the anterior segment findings after non-penetrating deep sclerectomy and the filtering blebs of eyes that underwent glaucoma filtering surgery.

Patients scheduled for Ahmed Tube surgery, with or without lens extraction and intraocular lens implant, will be recruited and randomized into two groups. The first group of patients will have a pericardial patch graft covering the tube, and fibrin glue will be used to attach the graft to the sclera and to close the conjunctiva. The second group will have a partial- thickness scleral flap raised to cover the tube, and the conjunctiva will be closed with conventional sutures.

ELIGIBILITY:
Inclusion Criteria:

* More than 40 years old
* Able to give informed consent
* Diagnosis of any type of glaucoma needing a Glaucoma drainage device (Ahmed tube implant) with or without lens extraction and intraocular lens implant because of uncontrolled intraocular pressures inspite of maximum tolerated medical therapy

Exclusion Criteria:

* Inability to give informed consent
* History of ocular infection or inflammation in the past two months

Min Age: 41 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-02; Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
Anterior segment optical coherence tomography appearance and measurements of the overlying conjunctiva, areas above and beneath the pericardial patch graft or partial thickness scleral flap, anterior chamber depth
Intraocular pressure

CONTACTS AND LOCATIONS:
Overall Officials: Paul Chew, FRCSEd,MMed, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Savini G, Zanini M, Barboni P. Filtering blebs imaging by optical coherence tomography. Clin Exp Ophthalmol. 2005 Oct;33(5):483-9. doi: 10.1111/j.1442-9071.2005.01066.x. PMID 16181273
- [Background] Kahook MY, Noecker RJ. Fibrin glue-assisted glaucoma drainage device surgery. Br J Ophthalmol. 2006 Dec;90(12):1486-9. doi: 10.1136/bjo.2006.101253. Epub 2006 Aug 17. PMID 16916877